CLINICAL TRIAL: NCT03062540
Title: A Phase 3, Double-Blind, Randomized, Multicenter, Placebo-Controlled Study to Evaluate the Efficacy and Safety of TNX-102 SL Taken Daily at Bedtime in Patients With Military-Related PTSD
Brief Title: Safety and Efficacy Study of TNX-102 SL in Patients With Military-related PTSD
Acronym: HONOR
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Stopped early due to inadequate separation on primary efficacy endpoint at Week 12 according to Interim Analysis conducted on the first 274 (50%) patients.
Sponsor: Tonix Pharmaceuticals, Inc. (Industry)
Collaborators: Premier Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TNX-CY-P301
Record Dates: First submitted 2017-02-20; First posted 2017-02-23 (Actual); Results first posted 2024-05-22 (Actual); Last update posted 2024-05-22 (Actual); Status verified 2024-04

CONDITIONS: PTSD
Keywords: PTSD; Military-related PTSD
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- TNX-102 SL Tablet, 5.6 mg (Experimental): 2 x TNX-102 SL, 2.8 mg Tablets taken sublingually each day at bedtime for 12 weeks.
  Interventions: Drug: TNX-102 SL
- Placebo SL Tablet (Placebo Comparator): 2 x Placebo Tablet taken sublingually each day at bedtime for 12 weeks.
  Interventions: Drug: Placebo SL Tablet

INTERVENTIONS:
Drug: TNX-102 SL — Patients will take 2 tablets of randomly assigned study drug sublingually each day at bedtime starting on Day 0 for 12 weeks
  Other Names: Low dose cyclobenzaprine sublingual tablets
  Arms: TNX-102 SL Tablet, 5.6 mg
Drug: Placebo SL Tablet — Patients will take 2 tablets of randomly assigned study drug sublingually each day at bedtime starting on Day 0 for 12 weeks
  Other Names: Placebo sublingual tablets
  Arms: Placebo SL Tablet

SUMMARY:
This is a 12-week, multicenter, randomized, double-blind, placebo-controlled, fixed-dose study that will investigate the efficacy and safety of 5.6 mg TNX-102 SL (2 x 2.8 mg tablets)-a sublingual formulation of cyclobenzaprine. Following successful screening and randomization, eligible patients will have a telephonic visit at week 2 and then return regularly to the study clinic for monthly visits for assessments of efficacy and safety.

ELIGIBILITY:
Inclusion Criteria:

* Male or female between 18 and 75 years of age, who have served in any branch of the military.
* Diagnosed with current PTSD as determined by the Clinician-Administered PTSD Scale (CAPS-5) for DSM-5.
* Index trauma(s) resulting in PTSD must meet DSM-5 criterion A for PTSD as described in CAPS-5, have occurred in 2001 or later, be military service related.
* Willing to refrain from use of all other formulations of cyclobenzaprine.
* Willing and able to refrain from antidepressants and other excluded medications.
* Capable of reading and understanding English and able to provide written informed consent.
* If female, either not of childbearing potential or practicing a medically acceptable method of birth control throughout the study.
* Willing and able to comply with all protocol-specified requirements.

Exclusion Criteria:

* Increased risk of suicide, based on the investigator's judgment that is of a severity that is not appropriate for outpatient management, or that warrants additional therapy excluded by the protocol.
* Significant (e.g., moderate or severe) comorbid traumatic brain injury (TBI) by history.
* Severe depressive symptoms at screening or baseline.
* Clinically significant laboratory abnormalities based on screening laboratory tests and/or medical history in the investigator's opinion.
* Use of antidepressant medication within 2 months of baseline.
* Female patients who are pregnant or lactating.
* History of serotonin syndrome, severe allergic reaction or bronchospasm or known hypersensitivity to cyclobenzaprine or the excipients.
* Seizure disorder.
* Patients with a body mass index (BMI) > 45.
* Has received any other investigational drug within 30 days before Screening.
* Previous participation in any other study with TNX-102 SL.
* Family member of investigative staff.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 358 (Actual)
Dates: Start 2017-03-27 (Actual); Primary Completion 2018-07-27 (Actual); Study Completion 2018-07-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Greg Sullivan, MD, Study Director — Tonix Pharmaceuticals
Locations (43):
- United States (43):
  - Phoenix, Phoenix, Arizona
  - Little Rock, Little Rock, Arkansas
  - Rogers, Rogers, Arkansas
  - Beverly hills, Beverly Hills, California
  - Glendale, Glendale, California
  - Oakland, Oakland, California
  - Oceanside, Oceanside, California
  - Orange, Orange, California
  - Riverside, Riverside, California
  - San Diego, San Diego, California
  - Temecula, Temecula, California
  - Colorado Springs, Colorado Springs, Colorado
  - Cromwell, Cromwell, Connecticut
  - Norwich, Norwich, Connecticut
  - Washington, D.C., Washington D.C., District of Columbia
  - Jacksonville, Jacksonville, Florida
  - Lake City, Lake City, Florida
  - Lauderhill, Lauderhill, Florida
  - Maitland, Maitland, Florida
  - Tampa, Tampa, Florida
  - Atlanta, Atlanta, Georgia
  - Chicago, Chicago, Illinois
  - New Bedford, New Bedford, Massachusetts
  - Flowood, Flowood, Mississippi
  - St. Louis, St Louis, Missouri
  - Missoula, Missoula, Montana
  - Las Vegas, Las Vegas, Nevada
  - Berlin, Berlin, New Jersey
  - Cedarhurst, Cedarhurst, New York
  - New York, New York, New York
  - Canton, Canton, Ohio
  - Cincinnati, Cincinnati, Ohio
  - Dayton, Dayton, Ohio
  - Oklahoma City, Oklahoma City, Oklahoma
  - Downingtown, Downingtown, Pennsylvania
  - Media, Media, Pennsylvania
  - Charleston, Charleston, South Carolina
  - Austin, Austin, Texas
  - Dallas, Dallas, Texas
  - Houston, Houston, Texas
  - San Antonio, San Antonio, Texas
  - Salem, Salem, Virginia
  - Everett, Everett, Washington

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Parmenter ME, Lederman S, Weathers FW, Davis LL, Vaughn B, Engels J, Sullivan GM. A phase 3, randomized, placebo-controlled, trial to evaluate the efficacy and safety of bedtime sublingual cyclobenzaprine (TNX-102 SL) in military-related posttraumatic stress disorder. Psychiatry Res. 2024 Apr;334:115764. doi: 10.1016/j.psychres.2024.115764. Epub 2024 Feb 1. PMID 38350291
- [Derived] Dunlop BW, Rakofsky JJ, Newport DJ, Mletzko-Crowe T, Barone K, Nemeroff CB, Harvey PD. Efficacy of Vortioxetine Monotherapy for Posttraumatic Stress Disorder: A Randomized, Placebo-Controlled Trial. J Clin Psychopharmacol. 2021 Mar-Apr 01;41(2):172-179. doi: 10.1097/JCP.0000000000001363. PMID 33587394

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | TNX-102 SL Tablet, 5.6 mg | Placebo SL Tablet
Started | 179 | 179
Completed | 110 | 120
Not Completed | 69 | 59

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | TNX-102 SL Tablet, 5.6 mg | Placebo SL Tablet | Total
Number analyzed (Participants) | 179 | 179 | 358
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.4 (8.21) | 35.9 (7.69) | 35.7 (7.95)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 21 | 36
  Male | 164 | 158 | 322
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 35 | 34 | 69
  Not Hispanic or Latino | 144 | 145 | 289
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 4 | 4 | 8
  Asian | 7 | 6 | 13
  Native Hawaiian or Other Pacific Islander | 4 | 3 | 7
  Black or African American | 31 | 31 | 62
  White | 122 | 124 | 246
  More than one race | 4 | 6 | 10
  Unknown or Not Reported | 7 | 5 | 12
Region of Enrollment [Number; unit: participants]
  United States | 179 | 179 | 358

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline in the Total Clinician Administered PTSD Scale (CAPS-5) for DSM-5 at Week 12.
Description: To evaluate the efficacy of the TNX-102 SL (cyclobenzaprine HCl sublingual tablets) using the Clinician Administered PTSD Scale for Diagnostic and Statistical Manual of Mental Disorders (DSM-5) (CAPS-5) total symptom severity score in a 12-week study. Score ranges from 0 to 80 with lower scores indicating less severe PTSD symptoms.
Time Frame: Day 0 and Week 12
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | TNX-102 SL Tablet, 5.6 mg | Placebo SL Tablet
Number analyzed (Participants) | 125 | 127
units on a scale | -15.2 (1.90) | -14.2 (1.80)

2. Secondary Outcome: Clinical Global Impression - Improvement From Initiation of Treatment (CGI-I) Score After 12 Weeks of Treatment.
Description: To evaluate the efficacy of the TNX-102 SL (cyclobenzaprine HCl sublingual tablets) using the CGI-I score after 12 weeks of treatment. Score ranges from 1 to 7. 1 = Very much improved. 2 = Much improved. 3 = Minimally improved. 4 = No change. 5 = Minimally worse. 6 = Much worse. 7 = Very much worse.
Time Frame: Week 12
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | TNX-102 SL Tablet, 5.6 mg | Placebo SL Tablet
Number analyzed (Participants) | 100 | 106
score on a scale | 2.6 (0.16) | 2.7 (0.15)

3. Secondary Outcome: Change From Baseline in the Disruption of Social Life/Leisure Activities Assessed Using the Sheehan Disability Scale (SDS) After 12 Weeks of Treatment.
Description: To evaluate the efficacy of the TNX-102 SL (cyclobenzaprine HCl sublingual tablets) using the change from baseline in disruption of social life/leisure activities assessed with the SDS after 12 weeks of treatment. Score ranges from 0 to 10. Lower scores indicate less disruption to social life/leisure activities.
Time Frame: Day 0, Week 12.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | TNX-102 SL Tablet, 5.6 mg | Placebo SL Tablet
Number analyzed (Participants) | 100 | 106
units on a scale | -2.1 (0.38) | -1.7 (0.35)

4. Secondary Outcome: Change From Baseline in the Disruption of Work/School Activities Assessed Using the Sheehan Disability Scale (SDS) After 12 Weeks of Treatment.
Description: To evaluate the efficacy of the TNX-102 SL (cyclobenzaprine HCl sublingual tablets) using the change from baseline in disruption of work/school activities assessed with the SDS after 12 weeks of treatment. Score ranges from 0 to 10. Lowers scores indicate less disruption to work/school activities.
Time Frame: Day 0, Week 12.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | TNX-102 SL Tablet, 5.6 mg | Placebo SL Tablet
Number analyzed (Participants) | 77 | 84
units on a scale | -1.6 (0.46) | -1.3 (0.41)

5. Secondary Outcome: Change From Baseline in Patients' Quality of Sleep Using the Patient-Reported Outcome Measurement Information System (PROMIS) Sleep Disturbance Scale After 12 Weeks of Treatment.
Description: To evaluate the efficacy of the TNX-102 SL (cyclobenzaprine HCl sublingual tablets) using the change from baseline in quality of sleep using the PROMIS Sleep Disturbance scale after 12 weeks of treatment. Raw score is transformed to T-scores using published conversions. T-score ranges from 30 to 80 with lower scores indicating better sleep quality.
Time Frame: Day 0, Week 12.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | TNX-102 SL Tablet, 5.6 mg | Placebo SL Tablet
Number analyzed (Participants) | 100 | 105
units on a scale | -9.3 (1.60) | -6.7 (1.49)

ADVERSE EVENTS:
Time Frame: 12 weeks
Description: The denominator used for calculating adverse event frequencies was the number of patients confirmed to have taken at least one dose of study medication. Therefore, the denominator used for calculating the frequency differs from the total number of enrolled patients.
  All-cause mortality was calculated using all patients as the denominator.
Arm/Group | TNX-102 SL Tablet, 5.6 mg | Placebo SL Tablet
All-Cause Mortality (participants affected / at risk) | 0/179 | 0/179
Serious Adverse Events (participants affected / at risk) | 3/175 | 5/176
Other Adverse Events (participants affected / at risk) | 93/175 | 21/176
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | TNX-102 SL Tablet, 5.6 mg (N=175) | Placebo SL Tablet (N=176)
Suicidal Ideation (Psychiatric disorders) | 1 | 1
Alcohol Withdrawal Syndrome (Psychiatric disorders) | 1 | 0
Suicide Attempt (Psychiatric disorders) | 0 | 1
Amaurosis fugax (Eye disorders) | 0 | 1
Cholangitis (Hepatobiliary disorders) | 0 | 1
Femur Fracture (Injury, poisoning and procedural complications) | 1 | 0
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | TNX-102 SL Tablet, 5.6 mg (N=175) | Placebo SL Tablet (N=176)
Hypoaesthesia Oral (Gastrointestinal disorders) | 70 | 2
Paraesthesia Oral (Gastrointestinal disorders) | 16 | 1
Somnolence (Nervous system disorders) | 27 | 15
Product Taste Abnormal (Product Issues) | 17 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
An industry standard NDA is in place with all study investigators.

DOCUMENTS (2):
  • Study Protocol (2019-10-29): https://cdn.clinicaltrials.gov/large-docs/40/NCT03062540/Prot_000.pdf
  • Statistical Analysis Plan (2018-05-16): https://cdn.clinicaltrials.gov/large-docs/40/NCT03062540/SAP_001.pdf